CLINICAL TRIAL: NCT05909215
Title: Attenuation Of Hemodynamic Response To Laryngoscopy. Role Of Dexmedetomidine. A Dose Finding Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sindh Institute of Urology and Transplantation (Other)
Responsible Party: Principal Investigator, Syed Muhammad Abbas, Associate Professor, Department of Anaesthesia, Sindh Institute of Urology and Transplantation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SindhInstitute
Record Dates: First submitted 2023-02-07; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Hemodynamic Instability; Tracheal Intubation; Dexmedetomidine
Keywords: Systolic Blood Pressure; Diastolic Blood Pressure; Heart Rate; Mean Arterial Pressure; Precedex; Tracheal Intubation; Laryngoscopy; Sedation
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dexmedetomidine 0.5 (Active Comparator): Dexmedetomidine 0.5 μ/kg diluted in 20 mL normal saline through a syringe pump over 10 minutes followed by general anesthesia.
  Interventions: Drug: Normal saline; Drug: Dexmedetomidine 0.5 microgram/kg
- Dexmedetomidine 0.75 (Active Comparator): Dexmedetomidine 0.75 μ/kg diluted in 20 mL normal saline through a syringe pump over 10 minutes followed by general anesthesia.
  Interventions: Drug: Normal saline; Drug: Dexmedetomidine 0.75 microgram/kg
- Placebo (Placebo Comparator): 20 mL of normal saline as an infusion through a syringe pump over 10 minutes followed by induction of general anesthesia.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Normal saline — Normal saline 20mL will be given intravenously through a syringe pump over 10 minutes
  Other Names: Placebo group
Drug: Dexmedetomidine 0.5 microgram/kg — Dexmedetomidine 0.5 microgram/kg diluted in 20mL of normal saline will be given intravenously through a syringe pump over 10 minutes
  Arms: Dexmedetomidine 0.5
Drug: Dexmedetomidine 0.75 microgram/kg — Dexmedetomidine 0.75 microgram/kg diluted in 20mL of normal saline will be given intravenously through a syringe pump over 10 minutes
  Arms: Dexmedetomidine 0.75

SUMMARY:
Two doses of Dexmedetomidine (0.5 µ/kg and 0.75 µ/kg) will be used to attenuate the stress response to laryngoscopy in American Society of Anesthesiology, physical class I patients which will be compared with the placebo-controlled group.

DETAILED DESCRIPTION:
A randomized, double-blind controlled trial will be conducted to determine the attenuation of stress response caused by laryngoscopy and tracheal intubation (LTI). After the Institutional Ethics Committee approval, (Sindh Institute of Urology and Transplantation, Pakistan), written informed consent will be obtained from 105 adult patients.

Randomization will be done using a computer-generated random number table. Patients will be divided into three groups. Group A "Placebo group", will receive 20 mL of normal saline (NS), Group B "dexmedetomidine 0.5", will receive dexmedetomidine 0.5 μ/kg, whereas, Group C "dexmedetomidine 0.75", will receive dexmedetomidine 0.75 μ/kg, all as a 20mL infusion through a syringe pump over 10 minutes followed by induction of general anesthesia.

No premedication will be given in the ward. Once the patients will arrive in the operating room, routine monitoring (electrocardiogram, pulse oximetry, non-invasive blood pressure) will be started. After recording the baseline vitals and Ramsay sedation score, the study drug or normal saline (according to randomization) will be given in a look-alike syringe over 10 minutes. The study drug will be prepared as a 20 mL solution in a 25 mL syringe. An independent co-investigator (anaesthesiologist) who will not be involved in administering general anesthesia or recording the study parameters will prepare the study drug(s) according to the body weight or NS using identical-looking syringes. Study drug infusion will be started once the patient is taken to the operating table. Vitals and sedation scores will be recorded at 0,1,3,5 and 10 minutes during infusion. Investigators will keep the atropine drawn in a syringe and ready to be given in case of heart rate goes below 40 beats/min. Ephedrine (5mg/ml) and adrenaline 10µ/ml will also be ready for use.

Once completing the infusion, general anesthesia will be administered using a standard protocol (Nalbuphine 0.15 mg/kg, Propofol 2.5 mg/kg, Atracurium 0.6 mg/kg after assessing easy bag-mask ventilation in all patients. After 3-minute bag-mask ventilation with Isoflurane at 1.5% in 100% oxygen, the trachea will be intubated by one of three senior anaesthesiologists involved in this study. The intubating duration will be kept below 15 seconds. Hemodynamic monitoring will be continued for another 10 minutes at 1, 3, 5 and 10 minutes after intubating the trachea.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 55 years
* ASA I or II patients undergoing surgery under general anaesthesia with endotracheal intubation.
* Patients with Mallampati class I or II.

Exclusion Criteria:

* ASA III & IV patients
* Anticipated or unanticipated difficult intubations which requires more than 15 seconds or more than one attempt.
* Patients with Mallampati class III, IV or with loose teeth.
* Patients with inotropes infusion.
* Patients with known allergy to any anaesthetic agents
* Patients with a heart rate of 60 beats/min or less
* Patients with known hypertension, incidental finding of hypertension while on operating table, diabetes, ischemic heart disease or peripheral vascular disease.
* Pregnant and lactating mothers.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Hemodynamic Response | 0 to 10 minutes after endotracheal intubation
  Mean change in the heart rate, systolic blood pressure, diastolic blood pressure, and mean arterial pressure will be assessed.

SECONDARY OUTCOMES:
Adverse events | 0 to 30 minutes from the start of infusion to 10 minutes after endotracheal intubation)
  Adverse events after intervention such as drowsiness, nausea, vomiting, or severe bradycardia will be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Syed M Abbas, Principal Investigator — Associate Professor Dept of Anaesthesia
Locations (1):
- Syed Muhammad Abbas, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No